CLINICAL TRIAL: NCT00124813
Title: Thalidomide, Cyclophosphamide, Oral Idarubicin and Dexamethasone (T-CID) as Induction Therapy and a Randomized Trial of Thalidomide vs Thalidomide Plus Oral Idarubicin as Maintenance Therapy in Patients With Multiple Myeloma
Brief Title: Thalidomide, Cyclophosphamide, Oral Idarubicin and Dexamethasone (T-CID) in Patients With Multiple Myeloma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Prof. Dr. I. Schmidt-Wolf, University Hospital, Bonn, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T-CID
Record Dates: First submitted 2005-07-27; First posted 2005-07-28 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Thalidomide; Idarubicin

INTERVENTIONS:
Drug: thalidomide
Drug: idarubicin — oral idarubicin

SUMMARY:
Background: In some studies, thalidomide in combination with chemotherapy has been shown to be effective in patients with relapsed or refractory multiple myeloma (MM). In this study, the researchers have chosen a regimen which can be administered on an outpatient basis.

Induction therapy: To evaluate the efficacy and toxicity of thalidomide, cyclophosphamide, oral idarubicin and dexamethasone (T-CID) in patients with relapsed or refractory multiple myeloma.

Maintenance therapy: Randomized trial to compare efficacy and toxicity of thalidomide and thalidomide plus oral idarubicin as maintenance therapy in patients with at least stable disease after T-CID.

DETAILED DESCRIPTION:
Background: In some studies, thalidomide in combination with chemotherapy has been shown to be effective in patients with relapsed or refractory multiple myeloma (MM). In this study, the researchers have chosen a regimen which can be administered on an outpatient basis.

After 3-8 cycles of T-CID patients with at least stable disease will be randomized to receive thalidomide or thalidomide plus oral idarubicin as maintenance therapy for at least one year or until progression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple myeloma according to British Columbia Cancer Agency Criteria
* Stage IIA/B or IIIA/B according to Durie/Salmon
* Symptomatic or progressive disease
* Status of disease:

  * refractory disease after standard induction therapy
  * OR relapse after standard induction therapy
  * OR relapse after high-dose chemotherapy/stem cell transplantation
  * OR patients with plasma cell leukemia
* Patients with measurable paraprotein in urine or serum or quantifiable bone marrow infiltration
* Written informed consent

Exclusion Criteria:

* Age < 18 years
* Life expectancy of less than 3 months
* Intolerance to the study drugs
* No change or progressive disease after prior therapy with idarubicin or cyclophosphamide
* Cardiac insufficiency New York Heart Association (NYHA) grade 3 or 4
* Acute infection
* Actually decompensated diabetes mellitus
* Total bilirubin > 3.0 mg/dl
* Pregnant or breast-feeding women
* Polyneuropathy grade 2 or higher
* Ulcus ventriculi or duodeni
* Narrow or open angle glaucoma
* Not-compensated psychiatric diseases
* Prior erythroblastopenia
* Prior therapy with investigational drugs within the last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2002-08; Primary Completion 2010-05 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Induction therapy: response rate, overall survival, death rate
Maintenance therapy: progression-free survival, overall survival, number of patients discontinuing therapy due to toxicity

SECONDARY OUTCOMES:
Induction therapy: number of patients discontinuing therapy due to toxicity, number of patients experiencing toxicity grade 3 or 4
Maintenance therapy: dose intensity, number of patients experiencing toxicity grade 3 or 4

CONTACTS AND LOCATIONS:
Overall Officials: Ingo Schmidt-Wolf, MD, Principal Investigator — University of Bonn
Locations (1):
- Medical Clinic & Policlinic III, University of Bonn, Bonn, Germany

REFERENCES:
- See also: Related Info — http://www.myelom.net